CLINICAL TRIAL: NCT06017505
Title: Integrating the Electronic Self-administered Gerocognitive Examination (eSAGE) With Electronic Health Records (EHR) Data Using Machine Learning (ML) for the Early Detection and Monitoring of Cognitive Impairment in Individuals
Brief Title: Integrating eSAGE With EHR Data Using Machine Learning for the Early Detection and Monitoring of Cognitive Impairment in Individuals
Status: Enrolling by invitation | Type: Observational
Sponsor: Douglas Scharre (Other)
Responsible Party: Sponsor-Investigator, Douglas Scharre, Professor-Clinical, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2023H0249
Record Dates: First submitted 2023-08-15; First posted 2023-08-30 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Dementia; Alzheimer Disease; Mild Cognitive Impairment; Worried Well
MeSH Terms: conditions — Dementia; Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subject population: Males and females 50 years of age and over who complete the eSAGE as part of their office visit at the Center for Cognitive and Memory Disorders.
  Interventions: Diagnostic Test: electronic self administered gerocognitive examination (eSAGE)

INTERVENTIONS:
Diagnostic Test: electronic self administered gerocognitive examination (eSAGE) — A self-administered digital assessment that evaluates multiple cognitive domains: orientation, language, memory, executive function, calculations, abstraction, and visuospatial abilities, through multiple questions. Additionally, it includes the collection of six clinical variables: education, gender, race, family history of dementia, stroke, and emotion.

SUMMARY:
The goal of this observational trial is to leverage the electronic Self-Administered Gerocognitive Examination (eSAGE), a variety of metadata (a set of data that describes and gives information about other data) collected during eSAGE testing, electronic health records (EHR) information, and advanced machine learning (ML) techniques to develop a new tool that can aid in early-stage prediction of individuals with cognitive impairments.

DETAILED DESCRIPTION:
This is a retrospective and prospective record review trial for patients who are followed at the Center for Cognitive and Memory Disorders.

eSAGE assessment data (including cognitive data, behavioral data, timing data and other metadata) as well as varying amount of electronic health records (EHR) data will be collected on all eligible subjects. Machine learning techniques with feature selection will identify important EHR variables to determine what may be useful for the prediction of cognitive impairment.

Based on the EHR analysis additional questions will be added to the eSAGE to make an enhanced eSAGE version (eSAGE+). The goal of the eSAGE+ is to facilitate the identification of cognition impairment, and ultimately have a translational impact on Alzheimer's disease (AD) identification and management.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males and females 50 years of age and over who complete the eSAGE as part of their office visit at the Center for Cognitive and Memory Disorders.

Exclusion Criteria:

* None

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include males and females 50 years of age and over who complete the eSAGE as part of their office visit at the Center for Cognitive and Memory Disorders.
Sampling Method: Probability Sample
Enrollment: 1486 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) for the ROC analysis in predicting subjects with cognitive impairment from cognitively normal subjects. | 1 day visit
  AUC ranges in value from 0 to 1

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Scharre, Principal Investigator — Ohio State University
Locations (1):
- Nicole Vrettos, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No